CLINICAL TRIAL: NCT06271434
Title: Krill Oil Supplementation and Its Effect on Intestinal Permeability Markers in Elite Rowers.
Brief Title: Effects of Krill Oil on Intestinal Integrity Markers in Elite Rowers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Olej z kryla/jelita
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-02

CONDITIONS: Endothelial Dysfunction
Keywords: endotoxin; gastrointestinal symtoms; gut permeability
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: All competitors will be randomly divided into two groups (double-blind):
  A. supplemented (n = 15), who will receive one capsule of a supplement called THYROX (Atlantic krill oil) four times a day.
  B. control (n = 15) receiving placebo. The supplementation period will be six weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented (Experimental): (n = 15), who will receive one capsule of a supplement called THYROX (Atlantic krill oil) four times a day. The daily content of krill oil is 2000 mg, including omega-3 fatty acids 350 mg, EPA - 240 mg, DHA - 110 mg, phospholipids - 800 mg, astaxanthin 200 mg.
  The supplementation period will be six weeks. Intervention: Drug: THYROX (Atlantic krill oil).
  Interventions: Dietary Supplement: THYROX (Atlantic krill oil
- Control (Experimental): receiving placebo Intervention: Drug: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: THYROX (Atlantic krill oil — The daily content of krill oil is 2000 mg, including omega-3 fatty acids 350 mg, EPA - 240 mg, DHA- 110 mg, phospholipids - 800 mg, astaxanthin 200 mg.
  Arms: Supplemented
Dietary Supplement: Placebo — The control capsules will be made of olive oil of equal size and color.
  Arms: Control

SUMMARY:
The study aims to check the influence of krill oil on markers of intestinal injury and intoxication.

Research group: the research will be conducted in a homogeneous group of professional rowers (N=30), all competitors qualified for the Polish Youth Rowing Team, aged 18 - 24. The sample size was confiremed in statistical analyses.

Rowing performance test will be conducted at the beginning and at the end of the training camp. Participants will perform a test on a rowing ergometer (Concept II, USA); each subject will have to cover a distance of 2000 m in the shortest possible time which is the distance starting in rowing competitions. The results of both tests will be considered in the selection for the championship team; therefore, athletes will be well motivated to perform both tests with maximum effort.

Hypotesis:

The krill oil will infleunce the gut barier integrity.

DETAILED DESCRIPTION:
All competitors will be randomly divided into two groups (double-blind):

A. supplemented (n = 15), who will receive one capsule of THYROX (Atlantic krill oil) four times a day.

B. control (n = 15) receiving placebo. The supplementation period will be six weeks.

Characteristic of the supplement:

THYROX (Atlantic krill oil). The daily recommended intake of krill oil is 2000 mg, which includes 350 mg of omega-3 fatty acids, 240 mg of EPA, 110 mg of DHA, 800 mg of phospholipids, and 200 mg of astaxanthin.

Placebo will be produced by MLB Bitrade Sp. z o.o., Poznan.

Measurement: The project contractors will measure all parameters using the available equipment in the ZWKF laboratory in Gorzów Wielkopolski and commercial assay kits.

Polyethylene clotting activator tubes (9 ml) will be centrifuged to separate the morphotic elements from the serum using a centrifuge (3000 rpm for 10 min). The serum will be pipetted into several Eppendorf tubes, then frozen (temp. -80 °C). All the following biochemical parameters will be determined from the extracted serum:

using the ELISA method by the test manufacturer's instructions. The designations include the flowing parameters:

a food diary will be filled day before the study and in the morning before the test, markers of gut injury: I-FABP (intestinal fatty acid binding protein), CLDN-3 (claudin 3) intoxication: LBP (lipopolysaccharide binding protein) stress hormones: ACTH and cortisol will be determined using the colourimetric method on the SPECTROstar Nano reader.

The lactate (La) concentration will be determined from the capillary blood immediately after collection using a commercially available kit (Diaglobal, Germany).

ELIGIBILITY:
Inclusion Criteria:

* training experience of a minimum of five years,
* minimum training time per week 240 minutes,
* all competitors qualified for the Polish Youth Rowing Team,
* completing a food diary,
* finishing 2000m ergometer test.

Exclusion Criteria:

* Probiotics, prebiotics and antibiotic therapy within the last three months,
* dietary regime,
* gastrointestinal diseases,
* lactose intolerance.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-23 (Estimated); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
I-FABP (intestinal fatty acid binding protein) | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  gut injury (enterocyte)
CLDN-3 | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  gut injury (tight junction)
LBP (lipopolysaccharide binding protein) | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  endotoxin
Catechyloamines, cortisol | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  stress hormones
CD14 | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  endotoxin

SECONDARY OUTCOMES:
Food intake | day before the test, morning before the test
  macro and micronutrients, fluids

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-S, professor, Study Director — Poznan University of Physical Education

IPD SHARING:
Plan to Share IPD: No